CLINICAL TRIAL: NCT02322697
Title: Effects of Chronic Intravenous Administration of L-carnitine on Myocardial Fatty Acid Metabolism in Hemodialysis Patients
Brief Title: Effect of Carnitine on Uremic Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toujinkai Hospital (Other)
Responsible Party: Principal Investigator, Masato Nishimura, MD, Director of cardiovascular division, Toujinkai Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dialysis heart carnitine study
Record Dates: First submitted 2014-10-08; First posted 2014-12-23 (Estimated); Last update posted 2014-12-25 (Estimated); Status verified 2014-12

CONDITIONS: Disorder of Fatty Acid Metabolism
Keywords: Carnitine; hemodialysis; fatty acid; imaging; heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carnitine group (Experimental): Intravenous administration of L-carnitine 1000mg after each hemodialysis session (three times a week) for one year.
  Interventions: Drug: Intravenous administration of L-carnitine
- control group (No Intervention): No intervention

INTERVENTIONS:
Drug: Intravenous administration of L-carnitine — Chronic intravenous administration of L-carnitine (1000mg on each dialysis session) for 1 year in hemodialysis patients
  Other Names: Chronic intravenous administration of L-carnitine
  Arms: Carnitine group

SUMMARY:
Patients on chronic hemodialysis without obstructive coronary artery disease identified by coronary angiography were randomly divided into the two groups: carnitine group and control group. SPECT using FFA analogue, BMIPP, was performed before and one year after intravenous administration of L-carnitine (1000 mg on every dialysis session). Control group received the examination of BMIPP SPECT at the same time of the carnitine group. The effects of chronic intravenous administration of L-carnitine on myocardial fatty acid metabolism were investigated among this population.

DETAILED DESCRIPTION:
Patients on chronic hemodialysis in Toujinkai hospital who had no obstructive coronary artery disease identified by coronary angiography and left ventricular dysfunction were randomly divided into the two groups: carnitine group and control group. To evaluate the possible effect of carnitine administration on myocardial fatty acid metabolism, SPECT using FFA analogue, BMIPP, was performed before and one year after intravenous administration of L-carnitine (1000 mg on every dialysis session). Control group received the examination of BMIPP SPECT at the same time of the carnitine group. Circulating concentrations of total, free, and acyl L-carnitine were measured every three months in the carnitine group. Clinical data including blood chemistry, blood pressure, or cardiac functions by echocardiography were obtained every 6 months in both groups. The effects of chronic intravenous administration of L-carnitine on myocardial fatty acid metabolism and cardiac functions were investigated among this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients on chronic hemodialysis without significant obstructive coronary artery disease identified by angiography within one years of the study, and who had left ventricular dysfunction:

  * reduced left ventricular systolic function (left ventricular ejection fraction <55%) and/or
  * left ventricular hypertrophy evaluated by echocardiography)

Exclusion Criteria:

1. Moderate or worse valvular heart disease,
2. Past histories of acute or old myocardial infarction and/or coronary revascularization by percutaneous coronary intervention or coronary artery bypass grafting within one year of the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
changes in BMIPP summed scores of the SPECT imaging | one year: September 2013-October 2014 (up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nishimura, MD, Principal Investigator — Toujinkai Hospital